CLINICAL TRIAL: NCT01275092
Title: CorPath® PRECISE Percutaneous Robotically-Enhanced Coronary Intervention Study (PRECISE)
Brief Title: Evaluation of the Safety and Effectiveness of the CorPath 200 System in Percutaneous Coronary Interventions (PCI)
Acronym: PRECISE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Corindus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CorPath PRECISE
Record Dates: First submitted 2011-01-07; First posted 2011-01-12 (Estimated); Results first posted 2013-08-08 (Estimated); Last update posted 2013-08-08 (Estimated); Status verified 2013-08

CONDITIONS: Coronary Artery Disease; Coronary Disease; Myocardial Ischemia; Heart Diseases; Cardiovascular Diseases; Arteriosclerosis; Arterial Occlusive Diseases; Vascular Diseases
Keywords: robotic-assisted PCI; coronary intervention; CorPath PRECISE; PCI
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease; Myocardial Ischemia; Heart Diseases; Cardiovascular Diseases; Arteriosclerosis; Arterial Occlusive Diseases; Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CorPath robotic-assisted PCI (Experimental): CorPath 200 robotic-assisted PCI
  Interventions: Device: CorPath robotic-assisted PCI

INTERVENTIONS:
Device: CorPath robotic-assisted PCI — CorPath 200® robotic-assisted percutaneous coronary intervention

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of the clinical and technical performance of the CorPath® 200 System in the delivery and manipulation of coronary guidewires and stent/balloon systems for use in percutaneous coronary interventions (PCI).

ELIGIBILITY:
General Inclusion Criteria:

1. Subject is between 18 and 99 years of age.
2. Subject is an acceptable candidate for PCI.
3. Subject must have clinical evidence of ischemic heart disease or a positive functional study.
4. Female subjects must be of non-child bearing potential, or if able to bear children, have a negative pregnancy test within 7 days prior to the CorPath procedure.
5. The subject or the legal representative has been informed of the nature of the study and agrees to its provisions and has provided written informed consent.

Angiographic Inclusion Criteria:

1. Study lesion is a single de novo native coronary artery lesion. This lesion may consist of multiple lesions (with 10mm or less between diseased segments) and must be completely covered by a single stent with at least 2.0mm of normal segments on proximal and distal edges of the lesion.
2. Study reference vessel diameter is between 2.5mm and 4.0mm by visual estimate.
3. Study lesion length is less than or equal to 24.0mm by visual estimate.
4. Study lesion diameter showing stenosis of at least 50% by visual estimate.

General Exclusion Criteria:

1. Subject requires planned PCI or CABG (Coronary Artery Bypass Graft) within 30 days following the CorPath procedure.
2. Evidence of an acute myocardial infarction within 72 hours prior to the intended CorPath procedure.
3. Subject has documented left ventricular ejection fraction <30%.
4. Subject has undergone PCI within 72 hours prior to the CorPath procedure.
5. Subject has undergone PCI within 30 days prior to the CorPath procedure and experienced a major adverse coronary event (MACE) or a serious adverse event (SAE) as defined in the protocol.
6. Subject has known hypersensitivity or contraindication to aspirin, heparin, ticlopidine, clopidogrel, prasugrel, stainless steel, cobalt chromium, or sensitivity to contrast media, including Visipaque™, which cannot be adequately pre-medicated or managed with clinically appropriate substitutes.
7. Subject has a platelet count <100,000 cells/mm3 or >700,000 cells/mm3, or a WBC (white blood cell) count of <3,000 cells/mm3 (e.g. thrombocytopenia, thrombocythemia, neutropenia or leukopenia).
8. Subject has a serum creatinine level of >2.0 mg/dL or eGFR (estimated Glomerular Filtration Rate) <30 ml/min as measured within 7 days prior to the procedure.
9. Subject has suffered a stroke within 30 days prior to planned CorPath procedure.
10. Subject has an active peptic ulcer or upper gastrointestinal bleeding within the 6 months prior to planned CorPath procedure.
11. Subject has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions.
12. Subject is currently participating in another investigational drug or drug/device or device trial and has not completed the entire follow up period.
13. Femoral access is not possible.

Angiographic Exclusion Criteria:

1. Target lesion that cannot be fully covered by a single stent.
2. Subject requires treatment of more than one vessel.
3. Any previous stent placement within 5.0 mm (proximal or distal) of the target lesion.
4. The study lesion requires planned treatment with directional coronary atherectomy (DCA), laser, rotational atherectomy or any device except for balloon dilatation prior to stent placement.
5. The study vessel has evidence of intraluminal thrombus.
6. The study vessel has evidence of moderate to severe tortuosity (>90°) proximal to the target lesion.
7. The study lesion has any of the following characteristics:

   * Total occlusion.
   * Ostial location.
   * Is within 2.0 mm of a side branch measuring >2.0 mm in diameter.
   * Located at < 45° bend in the vessel.
   * Moderately to severely calcified.
   * Moderate to severe calcification in the vessel proximal to the target lesion.
   * Located in a native vessel distal to an anastomosis, with a saphenous vein graft or a left/right internal mammary artery (LIMA/RIMA) bypass, and is approached through the bypass graft.
8. Unprotected left main coronary artery disease defined as an obstruction greater than 50% diameter stenosis in the left main coronary artery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michail Pankratov, MD/PhD, Study Director — Corindus Inc.
Locations (9):
- United States (8):
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Northeast Georgia Heart Center, Gainesville, Georgia
  - St. Elizabeth's Medical Center, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - Saint Joseph's Hospital, Syracuse, New York
  - Wellmont CVA Heart Institute, Kingsport, Tennessee
  - Virginia Commonwealth University, Richmond, Virginia
  - Swedish Medical Center, Seattle, Washington
- CORBIC, Medellín, Colombia

REFERENCES:
- [Derived] Weisz G, Metzger DC, Caputo RP, Delgado JA, Marshall JJ, Vetrovec GW, Reisman M, Waksman R, Granada JF, Novack V, Moses JW, Carrozza JP. Safety and feasibility of robotic percutaneous coronary intervention: PRECISE (Percutaneous Robotically-Enhanced Coronary Intervention) Study. J Am Coll Cardiol. 2013 Apr 16;61(15):1596-600. doi: 10.1016/j.jacc.2012.12.045. PMID 23500318

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During January-December 2011 period 164 participants were enrolled in the PRECISE study at 9 clinical sites
Period: Overall Study
Arm/Group | CorPath Robotic-assisted PCI
Started | 164
Completed | 164
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CorPath Robotic-assisted PCI
Number analyzed (Participants) | 164
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 87
  >=65 years | 77
Age Continuous [Mean (Standard Deviation); unit: years] | 64.1 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 122
Region of Enrollment [Number; unit: participants]
  United States | 144
  Colombia | 20

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinical Procedural Success
Description: Defined as <30% residual stenosis in CorPath 200 System treated lesions at the completion of the interventional procedure (including stent placement) in the absence of MACE, either within 48 hours of the procedure or prior to hospital discharge, whichever occurs first.
Time Frame: 48-hrs or hospital discharge, whichever occurs first
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CorPath Robotic-assisted PCI
Number analyzed (Participants) | 164
percentage of participants | 97.6 [94.5 to 100]

2. Primary Outcome: Percentage of Patients With Device Technical Success
Description: Defined as the successful advancement and retraction of PCI devices using the CorPath 200 System and without conversion to manual operation.
Time Frame: 1 day
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CorPath Robotic-assisted PCI
Number analyzed (Participants) | 164
percentage of participants | 98.8 [96.2 to 100]

3. Secondary Outcome: The Ratio Between the Radiation Exposure of the Primary Operator and the Radiation Exposure at the Table
Description: Defined as the difference between the radiation exposure measured at the procedure table (the conventional site of the primary operator) and the radiation exposure measured at the primary operator's position during the procedure. The radiation unit that was used was in milligray, but the measure is being reported as the ratio.
Time Frame: 1 day
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | CorPath Robotic-assisted PCI
Number analyzed (Participants) | 164
ratio | 0.42 [0 to 4.5]

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | CorPath Robotic-assisted PCI
Serious Adverse Events (participants affected / at risk) | 28/164
Other Adverse Events (participants affected / at risk) | 62/164
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CorPath Robotic-assisted PCI (N=164)
cardiovascular complications (Vascular disorders) | 27 (28)
Others (General disorders) | 1 (5)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CorPath Robotic-assisted PCI (N=164)
Cardiovascular complications (Vascular disorders) | 26 (26)
Others (General disorders) | 36 (36)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days